CLINICAL TRIAL: NCT00701974
Title: Study of Non Inferiority of Product Kollagenase ®, Manufactured by Laboratory Cristália When Compared With Iruxol ®, Manufactured by Abbott Laboratory, in the Treatment of Cutaneous Ulcers
Brief Title: Non-inferiority Clinic of Kollagenase® Compared Iruxol® in Treatment of Cutaneous Ulcers
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's strategy
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COLCRI0208; COLCRI0208 (Other: Protocol)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Ulcers
Keywords: Non-inferiority based on efficiency
MeSH Terms: conditions — Ulcer | interventions — Collagenases; iruxol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients treated with collagenase (IRUXOL)
  Interventions: Biological: collagenase (IRUXOL)
- 2 (Experimental): patients treated with collagenase (Kollagenase)
  Interventions: Biological: collagenase (Kollagenase)

INTERVENTIONS:
Biological: collagenase (IRUXOL) — patients will be treated with collagenase one time per day.
  Arms: 1
Biological: collagenase (Kollagenase) — patients will be treated with collagenase one time per day.
  Arms: 2

SUMMARY:
Skin ulcers can be defined as open injuries, loss of substances with the skin or mucous tissue, caused by disintegration and tissue necrosis. Chronic skin ulcer is any injury that heal in a period not less than 6 weeks. Several etiological causes for the emergence of skin ulcers. Around 73% are venous, arterial are 8%, 3% are diabetic, 2% are traumatic and 14% are from other causes.

Clinical studies show that collagenase is an effective drug and presents high tolerabildade in the treatment of ulcerative burns and injuries of various etiologies. Evidence show statistically significant reduction of inflammation, the formation of granulation tissue, decrease in injuries and reepitelization.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged over 18 years
* people with skin ulcers of the lower limbs for at least 3 months

Exclusion Criteria:

* Lesion with a diameter larger than 12 cm ²
* injury over 2 years of evolution; injury infected
* neoplastic lesions in activity
* poorly controlled diabetes mellitus
* HAS poorly controlled
* signs of ischemia in the limb
* not offset any disease
* allergic to components of formula
* urticaria
* pregnancy
* breastfeeding
* emotional disturbance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2008-02 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02

PRIMARY OUTCOMES:
Primary: Non-inferiority based on efficiency that will be evaluated by the general improvement of the injury; Secondary: tolerability assessed by the incidence of adverse events. | healing

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica, Valinhos, São Paulo, Brazil